CLINICAL TRIAL: NCT01411254
Title: A Randomized, Multicenter, Sham Controlled, Double-Masked, Phase 2/3 Study Assessing Efficacy and Safety of Betamethasone Microsphere in Patients With Diabetic Macular Edema
Brief Title: Efficacy and Safety of Betamethasone Microsphere in Patients With Diabetic Macular Edema (TSUBASA)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Other Study IDs: 01021103
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Diabetic Macular Edema
Keywords: DME
MeSH Terms: interventions — salicylhydroxamic acid

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Betamethasone Microsphere (DE-102） Low Dose
- 2 (Experimental)
  Interventions: Drug: Betamethasone Microsphere (DE-102） High Dose
- 3 (Sham Comparator)
  Interventions: Drug: Sham

INTERVENTIONS:
Drug: Betamethasone Microsphere (DE-102） Low Dose
  Arms: 1
Drug: Betamethasone Microsphere (DE-102） High Dose
  Arms: 2
Drug: Sham
  Arms: 3

SUMMARY:
This study will evaluate the efficacy and safety of Betamethasone Microsphere (DE-102) for diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed, written informed consent
* 20 years of age or older with diabetic macular edema

Exclusion Criteria:

* Active proliferative diabetic retinopathies (PDR) in the study eye
* Uncontrolled diabetes mellitus and hypertension
* Known steroid-responder

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Best Corrected Visual Acuity(BCVA)
  Change from baseline of Best Corrected Visual Acuity(BCVA) in ETDRS letter score

SECONDARY OUTCOMES:
retinal thickness
  Change in retinal thickness from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Santen study sites, Osaka, Osaka, Japan